CLINICAL TRIAL: NCT04332848
Title: Comparison of Susceptibility Testing Guided Versus Empirical Therapy for the Third-line Eradication of H. Pylori- a Multicenter Randomized Trial
Brief Title: Susceptibility Testing Guided Versus Empirical Therapy for Refractory H. Pylori Infection
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202001085MINB
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori,Susceptibility testing,empirical,third-line treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- (B) Empirical therapy (Experimental): choose antibiotics according to drug history
  Interventions: Drug: ET
- (A) Susceptibility testing guided therapy (Active Comparator): choose antibiotics according to susceptibility testing
  Interventions: Drug: SGT

INTERVENTIONS:
Drug: ET — Empirical therapy Based on drug history: Levofloxacin sequential therapy or bismuth quadruple therapy (10 or 14 days) or rifabutin triple/quadruple therapy or concomitant therapy
  Arms: (B) Empirical therapy
Drug: SGT — Susceptibility testing guided therapy Based on susceptibility test: Levofloxacin sequential therapy or bismuth quadruple therapy (10 or 14 days) or rifabutin triple/quadruple therapy or concomitant therapy
  Arms: (A) Susceptibility testing guided therapy

SUMMARY:
Aim: Therefore, we aimed to

1. compare the efficacy of susceptibility testing guided therapy vs. empirical therapy in the third-line eradication for refractory H. pylori infection
2. assess the long-term impact of eradication therapy on the antibiotic resistance and microbiota of the gut flora and the metabolic factors.

Methods: This will be a multi-center, open labeled trial

Patients: 360 patients with failure to H. pylori eradication for at least two times will be enrolled Determination of antibiotic resistance of H. pylori:

Agar dilution test will be used to determine the minimum inhibitory concentrations of levofloxacin, tetracycline, rifabutin, and clarithromycin to guide the selection of antibiotics.

Treatment regimens and assignment: Eligible patients will be randomized to receive either one of the treatments (A) Susceptibility testing guided therapy or (B) Empirical therapy

Outcome Measurement:

Primary End Point: Eradication rate will be evaluated according to Intent-to-treat (ITT) analyses.

Secondary End Point: 1. Eradication rate according to per protocol analysis (PP analysis); 2. Frequency of adverse effects.

ELIGIBILITY:
Inclusion criteria

* Adult (equal or greater than 20 years old) patients who failed from at least two eradication therapies for H. pylori infection will be enrolled.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2020-07-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the eradication rate in the third treatment according to intention-to treat (ITT) analysis. | 6 weeks
  Eradication rate will be determined by urea breath test at least 6 weeks after completion of treatment.

SECONDARY OUTCOMES:
Adverse effects | 2 weeks
  A standard interview and questionaire will be used to assess the adverse effects.

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Jyh Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan